CLINICAL TRIAL: NCT04496401
Title: Comparison of Pharmacokinetic (PK) Levels Before and After Conversion From Twice-daily Tacrolimus to Once-daily Extended-release Tacrolimus (LCPT) in Diabetic Transplant récipients
Brief Title: PK Study in Diabetic Transplant récipients : From Twice-daily Tacrolimus to Once-daily Extended-release Tacrolimus
Acronym: SPK-PK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC19_0247
Record Dates: First submitted 2020-07-23; First posted 2020-08-03 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-05

CONDITIONS: Kidney Transplantation; Pancreas Transplantation; Diabetes
Keywords: Tacrolimus; kidney transplant; pancreas transplant
MeSH Terms: conditions — Diabetes Mellitus | interventions — Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tacrolimus then Envarsus (Experimental): Tacrolimus will be started on the day of surgery. After a stable trough level is achieved (on postoperative day 7-17) the first PK profile will be measured. Subsequently, the switch to ENVARSUS® will be performed
  Interventions: Drug: Tacrolimus and Tacrolimus Extended Release Oral Tablet [Envarsus]

INTERVENTIONS:
Drug: Tacrolimus and Tacrolimus Extended Release Oral Tablet [Envarsus] — Phase 1: standard dose and frequency tacrolimus, used in accordance with licensing and local protocols. Suitable target trough level should be between 7-14 ng/ml.
  Phase 2: ENVARSUS® (LCP Tacro - extended release tacrolimus), used once-daily at an initial dose of 0.17mg/kg, dose adjusted to maintain an appropriate therapeutic blood concentration (measured by trough level). Suitable target trough level should be between 7-14 ng/ml.

SUMMARY:
The investigators believe that the pharmacological properties of Envarsus®, well studied in kidney transplantation, may be also suitable after simultaneous kidney and pancreas transplantation than Prograf. Indeed, Envarsus® has demonstrated a clinical efficacy and safety in a complete clinical development plan.

This study is to establish the pharmacokinetic profile of tacrolimus prolonged-release (hereafter referred to as 'ENVARSUS®') in diabetics who have undergone kidney and pancreas transplantation, and compare it to the pharmacokinetic profile of standard twice-daily tacrolimus. The study will be conducted in 25 patients hospitalized at Nantes University Hospital.

DETAILED DESCRIPTION:
The study will be conducted in 25 patients hospitalized at Nantes University Hospital. Tacrolimus will be started on the day of surgery (or on the day after) according to Nantes local standard doses and practices. After a stable trough level is achieved (on postoperative day 7-17) the first PK profile will be measured. Subsequently, the switch to ENVARSUS® will be performed (initial dose of 0.17 mg/kg/day) on a single morning oral dosage regimen. A second PK profile will be measured, between 7 to 14 days after initiation of ENVARSUS®. All these PK measurements will take place during the post-operative recovery in the hospital (typically 2-3 weeks). All patients will receive Thymoglobulin or Alemtuzumab induction, Myfortic or Cellcept (or generics), with or without prednisone according to local practices. Anti-infectious prophylaxis will be given according to Nantes local practices.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 18 years or above.
* Type I Diabetics patients with end stage chronic renal failure
* Recipient of kidney and pancreas-transplant
* At least one of the two transplants are functioning at time of PK profile measurements : a patient with early pancreatic graft failure due to thrombosis may be included if the kidney is well functioning
* Standard immunosuppressive therapy has been started post-operatively, in accordance with local policy, including tacrolimus.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Patients with social security.

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

* Patient is inappropriate for standard immunosuppressive therapy.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the patients at risk because of participation in the trial, or may influence the result of the trial, or the patient's ability to participate in the trial.
* Concomitant therapy with drugs potentially interfering with tacrolimus pharmacokinetics, especially those interfering with CYP3A4 (see 4.4 section in tacrolimus / ENVARSUS® summary of product characteristics).
* Loss of the pancreatic graft due to immunological causes
* Pregnant or breast-feeding women and female patient with potential childbearing refusing contraception.
* Vulnerable people: persons deprived of liberty; under trusteeship or under curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
To characterise the bioavailability of Envarsus® and compare it to the bioavailability of tacrolimus | Initial tacrolimus PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® PK profile measurement: day 15-32 post SPK transplantation
  To characterise the PK profile of extended release tacrolimus (Envarsus®) in diabetic transplant recipients, and compare it to the PK profile of tacrolimus : bioavailability AUC0-24

SECONDARY OUTCOMES:
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients with both functional grafts: Cmin | Initial tacrolimus and myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  Cmin
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients only with a functional kidney graft in case of early pancreas thrombosis.: Cmin | Initial tacrolimus and myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  Cmin
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients with both functional grafts : Cmax | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  Cmax
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients only with a functional kidney graft in case of early pancreas thrombosis.: Cmax | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  Cmax
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients with both functional grafts: Cavg | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  Cavg
Further quantification of the PK profile of extended release tacrolimus and Myforticin patients only with a functional kidney graft in case of early pancreas thrombosis.: Cavg | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  Cavg
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients with both functional grafts: Tmax | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  Tmax
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients only with a functional kidney graft in case of early pancreas thrombosis..: Tmax | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  Tmax
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients with both functional grafts : Ke | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  Ke
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients only with a functional kidney graft in case of early pancreas thrombosis.: Ke | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  Ke
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients with both functional grafts : t1/2 | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  t1/2
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients only with a functional kidney graft in case of early pancreas thrombosis.: t1/2 | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  t1/2
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients with both functional grafts: % fluctuation | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  % fluctuation
Further quantification of the PK profile of extended release tacrolimus and Myfortic in patients only with a functional kidney graft in case of early pancreas thrombosis: % fluctuation | Initial tacrolimus and Myfortic PK profile measurement: day 7-17 post SPK transplantation. Second ENVARSUS® and Myfortic PK profile measurement: day 15-32 post SPK transplantation
  % fluctuation
Assessment of biological and clinical tolerance/ safety: Incidence of serious adverse events | Months 6, or on leaving hospital if after 6 months (maximum one year after the inclusion)
  Incidence of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: DIEGO CANTAROVICH, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France